CLINICAL TRIAL: NCT02213653
Title: Phase IV Randomized Study Evaluating Agents Stimulants Erythropoiesis (ASE) Associated With Ferric Carboxymaltose (Ferinject ®) in Concomitant or Sequential Patients Treated for Cancer and With Anemia Associated With Functional Iron Deficiency
Brief Title: Randomized Study Evaluating Agents Stimulants Erythropoiesis (ASE) Associated With Ferric Carboxymaltose (Ferinject ®) in Concomitant or Sequential Patients Treated for Cancer and With Anemia Associated With Functional Iron Deficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry); Roche Pharma AG (Industry); Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FERASE
Record Dates: First submitted 2014-07-31; First posted 2014-08-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Solid Cancer Metastatic Disease; Lymphoid Disease
Keywords: Functional iron deficiency; Metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Concomitant iron and I.V. epoietin zeta (Experimental)
  Interventions: Drug: ARM A : IV iron + epoietin zeta
- Iron and I.V. epoietin zeta sequential (Experimental)
  Interventions: Drug: ARM B: IV iron + epoietin zeta sequence
- Epoietin zeta (Active Comparator)
  Interventions: Drug: ARM C : single epoietin zeta

INTERVENTIONS:
Drug: ARM A : IV iron + epoietin zeta — * Epoietin zeta at a dose of 450 IU / kg per week subcutaneously
  * Carboxymaltose ferric (Ferinject ®) at week 1; Intravenous infusion not exceeding 1000 mg (administered once if weight> 50 kg, 500 mg twice otherwise, with an interval of one week between each administration).
    * Renewable with a minimum of 4 weeks depending on the iron status (if CST <20% and absence of serum ferritin> 800) in the same manner as week 1.
  Arms: Concomitant iron and I.V. epoietin zeta
Drug: ARM B: IV iron + epoietin zeta sequence — * Epoietin zeta at a dose of 450 IU / kg per week subcutaneously started in week 7
  * carboxymaltose ferric (Ferinject ®) at week 1
    * Intravenous infusion not exceeding 1000 mg (administered once if weight> 50 kg, 500 mg twice otherwise, with an interval of one week between each administration).
    * Renewable with a minimum of 4 weeks depending on the iron status (if CST <20% and absence of serum ferritin> 800) in the same manner as week 1.
  Arms: Iron and I.V. epoietin zeta sequential
Drug: ARM C : single epoietin zeta — Epoietin zeta at a dose of 450 IU / kg per week subcutaneously begun in week 1
  Arms: Epoietin zeta

SUMMARY:
Anemia in patients with cancer is a common problem associated with an impaired quality of life.

Treatment with erythropoiesis stimulating agents (ESA) allows an increase in hemoglobin levels in 40-70% of patients and decreased transfusion requirements.

Absolute or functional iron deficiency is also common with about 30% of cancer patients with all histologies combined iron deficiency and anemia.

Several studies have shown the benefits of the combination of intravenous iron to erythropoiesis-stimulating agents in improving hemoglobin. However, none of them, to the investigators knowledge, has not been specifically performed on a population of patients with functional iron deficiency.

In addition, in clinical practice, this association is not carried out in particular because there is no dosage or consensus sequence for the administration of iron associated with ESAs.

DETAILED DESCRIPTION:
- Iron Deficiency and Cancer The literature review therefore presents uncertainties do not allow the routine application of intravenous iron associated with ESAs. The SOR also conclude that IV iron is "consider" if iron deficiency.

These uncertainties are the heterogeneity of the study populations, contradictory results and the use of patterns intravenous iron binding and non-standardized.

The investigators focus in this study in patients with chemotherapy-induced anemia with functional iron deficiency is a cause of lack of response to ESA. Indeed, patients with true iron deficiency seems to justify a routine iron supplementation. In contrast, patients without iron deficiency do not warrant formal way of initiating such treatment (although the literature is contradictory).

This study aims to evaluate, in patients with chemotherapy-induced anemia and functional iron deficiency, the efficacy and safety of the combination epoietin zeta + Iron in concomitant intravenous or sequential.

Because data RCP (Summary of Product Characteristics), ease of use, its safety profile, the ability to achieve higher doses of iron with a lower frequency and with better adherence, the ferric carboxymaltose was chosen as an intravenous iron. One specialty is available, the Ferinject ® (Laboratoires VIFOR Pharma).

The erythropoiesis-stimulating agent chosen in this study is epoietin zeta.

- Hepcidin and iron Hepcidin is a peptide hormone of 25 amino acids produced by the liver and considered as the central regulator of iron homeostasis in the body.

It works by controlling intestinal iron absorption and iron reuse by the reticuloendothelial system. Hepcidin acts by preventing the export of iron enterocytes, intestinal site of absorption of dietary iron, and macrophages, iron recycling site of hemoglobin, by binding to ferroportin present at the membrane these cells and by inducing its internalization and degradation.

Accordingly, hepcidin can be considered a hyposidérémiante hormone. The hepcidin rate is increased by the iron thereby limiting its accumulation and tissue damage associated with iron overload. Inversely, the rate is reduced hepcidin during increased iron as anemia needs, hypoxia, pregnancy or other situations of iron deficiency.

Moreover, hepcidin is strongly induced by inflammation. Thus, in pathological situations such as cancer, high levels of hepcidin explain well enough inflammatory anemia characterized by anemia, iron retention at storage proteins such as ferritin but also at the level of the reticuloendothelial system endothelial and a decrease in intestinal iron absorption.

Despite its importance in the pathophysiology of anemia of inflammation and a fortiori with iron deficiency anemia functional hepcidin is not measured in clinical routine. There is not, to the investigators knowledge, prospective data on its blood levels in situations of iron deficiency anemia in cancer patients functional and data on changes in hepcidin levels induced by treatment with intravenous iron or with erythropoietin.

ELIGIBILITY:
Inclusion Criteria:

* Patient> 18 years;
* Metastatic or locally advanced non-curable undergoing chemotherapy or lymphoid disease for which chemotherapy is indicated solid cancerous disease;
* Patient for which there are at least 3 cycles or 3 months of chemotherapy;
* Haemoglobin between 8.5 and 11 g / dL;
* Functional martial deficiency defined by a coefficient of transferrin saturation and serum ferritin ≤ 20% between 100 and 800 mg / L;
* Life expectancy> 3 months;
* ECOG ≤ 2.

Exclusion Criteria:

* Documented hemochromatosis ;
* AST and / or ALT> 2.5N;
* Renal impairment with Cockcroft clearance <30 mL / min;
* Vitamin B12 deficiency or folate;
* Hemolysis;
* Infectious disease being untreated;
* Haemorrhagic syndrome related or not with the tumor;
* Hypersensitivity to Ferinject ® or any of the excipients;
* Land atopic asthma or eczema known
* Contraindication to EPO;
* Taking a supplement to oral iron;
* Treatment with EPO within 6 months prior to study entry;
* No transfusion of packed red cells within 15 days before enrollment or randomization in the study;
* Participation in another clinical trial;
* Psychiatric pathology can disrupt the course of treatment or prevent the interpretation of results;
* Pregnant or lactating women;
* Persons deprived of liberty;
* Major subject to a measure of legal protection or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with hematopoietic response at 10 weeks. | The rate of hematopoietic response will be evaluated 10 weeks
  The primary objective is to evaluate the rate of hematopoietic response to 10 weeks in patients with anemia and functional iron deficiency treated epoietin zeta + carboxymaltose concomitant IV iron, by epoietin zeta + carboxymaltose IV ferric sequential or epoietin zeta alone

SECONDARY OUTCOMES:
Number of transfusion requirements | The number of transfusions will be evaluated weekly Week 1-16
  The secondary objective is to assess transfusion requirements will be evaluated throughout the study

OTHER OUTCOMES:
The hematopoietic response at 6 and 16 weeks | The hematopoietic response will be evaluated at 6 and 16 weeks
The time to achieve the therapeutic goal (hemoglobin> 12g/dl or increase in hemoglobin> 2g/dl) | The time to achieve the therapeutic goal will be determine 6,10 and 16 weeks after treatment start
Quality of life | Quality of life will be evaluated 6,10 and 16 weeks after treatment start
The consumption of erythropoiesis stimulating agent | The consumption of erythropoiesis stimulating agent will be evaluated 6,10 and 16 weeks after treatment start
The mean increase in hemoglobin concentration | The mean increase in hemoglobin concentration will be evaluated weekly Week 1-16
The evolution of the iron status parameters | The evolution of the iron status parameters will be performed at weeks 4,6,10,13 and 16
  Ferritin, CST, soluble transferrin receptor, reticulocytes, CRP will be dosed at weeks 4,6,10,13 and 16
Tolerance | Tolerance will be evaluated at weeks 6, 10 and 16
Fatigue | Fatigue will be evaluated 6,10 and 16 weeks after treatment start
  Fatigue will be estimated with the generic scale FACT-G

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel SEVIN, MD, Principal Investigator — Centre François Baclesse
Locations (2):
- France (2):
  - CHU, Caen
  - Centre François Baclesse, Caen